CLINICAL TRIAL: NCT05111431
Title: Study on Efficacy and Safety of Dexmedetomidine Hydrochloride Nasal Spray for Preoperative Sedation in Children
Brief Title: A Trial of Dexmedetomidine Hydrochloride Nasal Spray in Preoperative Sedation of Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HR0171401-302
Record Dates: First submitted 2021-10-20; First posted 2021-11-08 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2021-10

CONDITIONS: Preoperative Sedation of Children

STUDY DESIGN:
Intervention Model Description: Dexmedetomidine hydrochloride nasal spray compared with placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine Hydrochloride Nasal Spray (Experimental)
  Interventions: Drug: Dexmedetomidine Hydrochloride Nasal Spray
- Dexmedetomidine hydrochloride nasal spray blank preparation (Placebo Comparator)
  Interventions: Drug: Dexmedetomidine hydrochloride nasal spray blank preparation

INTERVENTIONS:
Drug: Dexmedetomidine Hydrochloride Nasal Spray — In the low weight group, the subjects will receive a low dose of dexmedetomidine nasal spray.
  In the high weight group, the subjects will receive a high dose of dexmedetomidine nasal spray.
  Arms: Dexmedetomidine Hydrochloride Nasal Spray
Drug: Dexmedetomidine hydrochloride nasal spray blank preparation — In the low weight group, the subjects will receive dexmedetomidine hydrochloride nasal spray blank preparation.
  In the high weight group, the subjects will receive dexmedetomidine hydrochloride nasal spray blank preparation.
  Arms: Dexmedetomidine hydrochloride nasal spray blank preparation

SUMMARY:
The study is being conducted to evaluate the efficacy, and safety of dexmedetomidine hydrochloride nasal spray for preoperative sedation in children.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide a written informed consent
2. Male or female
3. Subjects requiring elective general anesthesia surgery
4. Conform to the ASA Physical Status Classification
5. Meet the weight standard

Exclusion Criteria:

1. Not suitable for nasal spray
2. Pediatric populations requiring special care or court/social welfare supervision
3. Subjects who had been under general anesthesia when they were randomized
4. Subjects with a history of mental illness and a history of cognitive impairment epilepsy
5. Subjects with cardiovascular disease
6. Subjects whose hemoglobin is below the lower limit of normal
7. Subjects with a history or possibility of a difficult airway
8. Abnormal liver function and/or abnormal renal function
9. Adrenoceptor agonists or antagonists or analgesics were used before randomization
10. Participated in clinical trials (received experimental drugs)
11. History of hypersensitivity to drug ingredients or components
12. Other circumstances that the investigator judged inappropriate for participation in this clinical trial

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 159 (Actual)
Dates: Start 2021-11-24 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-05-20 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects who meet parent-child separation successful | within 45 minutes after the beginning of administration
Proportion of subjects who meet the Ramsay sedation score of 3 at least once within 45 minutes after the beginning of administration | within 45 minutes after the beginning of administration

SECONDARY OUTCOMES:
Proportion of subjects who meet parent-child separation successful within 45 minutes after the beginning of administration | Within 45 minutes after the beginning of administration
  The FUNK scale is a scale of 1 to 4 for sedation, anxiety, and separation from parents. Separation success is defined as a scale of 3 or 4 per item.
Time from the beginning of administration to the successful parent-child separation for the first time through study completion，an average of 3 days | an average of 3 days
  The FUNK scale is a scale of 1 to 4 for sedation, anxiety, and separation from parents. Separation success is defined as a scale of 3 or 4 per item.
Proportion of subjects whose the Ramsay score is satisfactory at least once within 45 minutes after the beginning of administration | Within 45 minutes after the beginning of administration
  Sedation level using the Ramsay scale. Ramsay Satisfaction is defined as a scale of ≥ 3.
Time from the beginning of administration to the satisfactory Ramsay score for the first time | from the beginning of administration to the first successful Ramsay score
  Sedation level using the Ramsay scale. Ramsay Satisfaction is defined as a scale of ≥ 3.
Proportion of subjects whose the UMSS Scale is satisfactory at least once within 45 minutes after the beginning of administration | within 45 minutes after the beginning of administration
  Sedation level using the University of Michigan Sedation Scale. UMSS satisfaction is defined as a scale of ≥ 2 .
Time from the beginning of administration to the satisfactory UMSS score for the first time through study completion，an average of 3 days | an average of 3 days
  Sedation level using the University of Michigan Sedation Scale. UMSS satisfaction is defined as a scale of ≥ 2.
Time of anesthesia awakening through study completion，an average of 3 days | an average of 3 days

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Children's Hospital Affiliated to Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gao J, Wang F, Wang X, Zou X, Liu HC, Song X, Chai X, Jiang R, Zhao P, Zhang J, Wang SY, Ma H, Zhao Z, Wang Q, Zhou N, Bai J, Zhang J. Safety and efficacy of a novel dexmedetomidine nasal spray for pre-anesthetic sedation in children: a randomized, double-blind, placebo-controlled trial. BMC Anesthesiol. 2024 Sep 6;24(1):315. doi: 10.1186/s12871-024-02708-1. PMID 39242499